CLINICAL TRIAL: NCT04008277
Title: Investigation of Heart Rate Variability During the Menstrual Cycle
Status: Completed | Type: Observational
Sponsor: SPD Development Company Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: PROTOCOL-1039
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Ovulation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Daily urine samples collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, women will be required to wear a heart rate monitor continuously and collect daily early morning urine samples for the duration of one complete menstrual cycle. This will enable comparisons between data collected from the heart rate monitor and hormone analysis in urine samples to be made.

DETAILED DESCRIPTION:
This pilot study is a prospective observational study of women's heart rate and heart rate variability throughout one complete menstrual cycle. A minimum of 10 volunteers aged 18 years of age or over will be recruited via a variety of methods according to the criteria detailed in section 9. They will be required to wear a heart rate monitor continuously and collect daily early morning urine samples throughout one menstrual cycle.

Urine samples will be returned to SPD on a regular basis for measurement of urinary hormones related to pregnancy and fertility. Data collected via the monitor including heart rate and heart rate variability will be downloaded for comparison.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and over
* Regular menstrual cycles

Exclusion Criteria:

* Taking any hormonal medications
* Taking any medications that may affect heart rate
* Known heart condition or use of a pacemaker
* Skin condition where there is sensitivity to wearing a skin monitor
* Currently suffering with anxiety or panic attacks
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2019-07-19 (Actual); Primary Completion 2019-10-02 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Heart Rate | 1 month
  Heart rate at time points throughout the menstrual cycle
Heart Rate Variability | 1 month
  Heart rate variability at time points throughout the menstrual cycle

SECONDARY OUTCOMES:
Day of ovulation | 1 month
  Day of ovulation determined by urinary LH surge +1 day
Fertile window | 1 month
  Fertile window onset determined by E3G surge
Fertile window closure | 1 month
  Fertile window closure determined by P3G rise

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Johnson, Study Director — SPD Development company Ltd.
Locations (1):
- SPD Development Company Ltd., Bedford, Bedfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No